CLINICAL TRIAL: NCT03271632
Title: Multiple Antigen-specific CAR T Cells For the Treatment of Multiple Myeloma
Brief Title: Multi-CAR T Cell Therapy in the Treatment of Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, Principal Investigator, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17013
Record Dates: First submitted 2017-08-27; First posted 2017-09-05 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; chimeric antigen receptor; BCMA; CD38; CD56; CD138
MeSH Terms: conditions — Multiple Myeloma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): CAR T cells to treat MM
  Interventions: Biological: CAR T cells

INTERVENTIONS:
Biological: CAR T cells — Infusion of multi-CAR T cells

SUMMARY:
The aim of this clinical trial is to assess the feasibility, safety and efficacy of autologous CAR T cell immunotherapy targeting multiple cancer cell surface antigens in relapsed and refractory multiple myeloma patients. Another goal of the study is to learn more about the persistence and function of CAR T cells in the body.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignancy of plasma cells, which remains a clinical challenge despite advanced therapeutic interventions including novel molecular therapies and stem cell transplantation (SCT). This trial is to test the safety and efficacy of T cells genetically modified to specifically target several MM surface antigens, including BCMA, CD38, CD56, CD138 or alternative MM surface antigens, based on a multi-CAR T cell immunotherapy approach. Another goal of the study is to investigate the persistence and function of CAR T cells in the body after CAR T cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with surface antigen confirmed multiple myeloma with no available curative treatment options (including autologous or allogeneic SCT).
* Complete remission (CR) cannot be achieved after at least 4 prior combination therapy regimens.
* MM in CR2 or CR3 and not eligible for allogeneic SCT because of age, comorbid diseases, or lack of available donor.
* Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval < 1 year).
* Relapsed after prior autologous or allogenic SCT MM patients with relapsed or residual disease after at least 1 prior therapy and not eligible for allogeneic SCT.
* Residual disease after primary therapy and not eligible for ASCT
* Expected survival > 12 weeks
* Creatinine < 2.5 mg/dl
* ALT (alanine aminotransferase)/AST (aspartate aminotransferase) < 3x normal
* Bilirubin < 2.0 mg/dl
* Any relapse after prior SCT is eligible regardless of other prior therapy
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given

Exclusion Criteria:

* Pregnant or lactating women
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Previous related CAR-T cell therapy Any uncontrolled active medical disorder that would preclude participation
* HIV infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with treatment related adverse effect | 1 month
  percentage of participants with treatment-related adverse events, as assessed by physical exam, vital signs, standard clinical lab tests.

SECONDARY OUTCOMES:
Anti-tumor activity of fourth generation multiple CAR-T cells after infusion | 1 year
  by measuring CAR copies in the body
Anti-tumor activity of fourth generation multiple CAR-T cells in patients with relapsed or refractory MM | 1 year
  by physical examination of tumor burden

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (2):
- China (2):
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - The First People's Hospital of Yunnan, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No